CLINICAL TRIAL: NCT02831179
Title: A Phase 1 Study of Veliparib (ABT-888) in Combination With Capecitabine and Temozolomide in Advanced Well-Differentiated Neuroendocrine Tumors
Brief Title: Veliparib, Capecitabine, and Temozolomide in Patients With Advanced, Metastatic, and Recurrent Neuroendocrine Tumor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding support
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jordan Berlin, MD, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 14134; NCI-2016-01044 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Functional Pancreatic Neuroendocrine Tumor; Malignant Somatostatinoma; Merkel Cell Carcinoma; Metastatic Adrenal Gland Pheochromocytoma; Metastatic Carcinoid Tumor; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2A; Multiple Endocrine Neoplasia Type 2B; Neuroendocrine Neoplasm; Non-Functional Pancreatic Neuroendocrine Tumor; Pancreatic Glucagonoma; Pancreatic Insulinoma; Recurrent Adrenal Cortex Carcinoma; Recurrent Adrenal Gland Pheochromocytoma; Recurrent Merkel Cell Carcinoma; Somatostatin-Producing Neuroendocrine Tumor; Stage III Adrenal Cortex Carcinoma; Stage III Thyroid Gland Medullary Carcinoma; Stage IIIA Merkel Cell Carcinoma; Stage IIIB Merkel Cell Carcinoma; Stage IV Adrenal Cortex Carcinoma; Stage IV Merkel Cell Carcinoma; Stage IVA Thyroid Gland Medullary Carcinoma; Stage IVB Thyroid Gland Medullary Carcinoma; Stage IVC Thyroid Gland Medullary Carcinoma; Thymic Carcinoid Tumor; VIP-Producing Neuroendocrine Tumor; Well Differentiated Adrenal Cortex Carcinoma; Zollinger Ellison Syndrome
MeSH Terms: conditions — Carcinoma, Merkel Cell; Pheochromocytoma; Carcinoid Tumor; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2a; Multiple Endocrine Neoplasia Type 2b; Neuroendocrine Tumors; Non functioning pancreatic endocrine tumor; Glucagonoma; Insulinoma; Adrenal Cortex Neoplasms; Somatostatinoma; Carcinoma, Medullary; Vipoma; Zollinger-Ellison Syndrome | interventions — Capecitabine; Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (capecitabine, temozolomide, veliparib) (Experimental): Capecitabine PO BID on days 1-14, temozolomide PO BID on days 10-14 and veliparib PO BID on days 10-14.
  Interventions: Drug: Capecitabine; Drug: Temozolomide; Drug: Veliparib; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Capecitabine — Given PO
Drug: Temozolomide — Given PI
Drug: Veliparib — given PO
Other: Pharmacological Study — Correlative studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with capecitabine and temozolomide in treating patients with neuroendocrine tumor that has spread to other places in the body and usually cannot be cured or controlled with treatment, has returned after a period of improvement, and cannot be removed by surgery. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of veliparib (ABT-888) in combination with capecitabine and temozolomide in patients with advanced well-differentiated neuroendocrine tumors.

SECONDARY OBJECTIVES:

2. To determine the safety profile of the combination of capecitabine, temozolomide and veliparib in patients with advanced well-differentiated neuroendocrine tumors (NET).

3. To evaluate the antitumor activity of the combination of capecitabine, temozolomide and veliparib in advanced well-differentiated NET patients

4. To determine progression-free survival (PFS) of the combination of capecitabine, temozolomide, and veliparib in advanced well-differentiated NET patients IV. To evaluate the association between pharmacodynamic biomarkers and response in patients with advanced well-differentiated NET patients.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive capecitabine orally (PO) twice daily (BID) on days 1-14, temozolomide PO BID on days 10-14 and veliparib PO BID on days 10-14. Courses repeat every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic unresectable well differentiated (low grade and intermediate grade) neuroendocrine tumors (Ki-67 < 20% and mitotic rate < 2 per 10 high power field) that demonstrate progressive disease (by serial computed tomography [CT] or magnetic resonance imaging [MRI] scans) in past 12 months including

  * Carcinoid tumors originating anywhere in the body including the gastrointestinal (GI) tract or bronchial tree or thymus
  * Pancreatic neuroendocrine tumors (including functional and non-functional islet cell, insulinomas and glucagonomas)
  * Pheochromocytomas
  * Gastrinomas (Zollinger-Ellison syndrome)
  * Multiple endocrine neoplasia (MEN type I/II),
  * Adrenal carcinomas with NET markers by immunohistochemistry (IHC) or serum
  * Somatostatinoma
  * VIPoma (vasoactive intestinal peptide)
  * Merkel cell tumors
  * Medullary thyroid carcinoma
  * Neuroendocrine tumors of unknown primary site
* Patients must have progressed on octreotide therapy and/or radioactive isotopes linked to octreotide or its congeners if they had a positive octreotide scan; patients who have negative or mildly positive octreotide scans are exempt from this requirement
* Somatostatin analogs can be continued at their tolerated dose in patients with functional symptoms related to underlying disease such as in functional islet cell, insulinomas, glucagonomas etc
* Patients may have received prior chemotherapy for advanced disease including either capecitabine or temozolomide single agent as long as it did not include combination of capecitabine and temozolomide
* Patients must have completed prior (non-excluded) anti-cancer therapy (including surgery or chemotherapy or hepatic embolization/chemoembolization or radioactive isotopes i.e. yttrium 90) at least 4 weeks prior to day 1
* Patients with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intracranial disease and have not had treatment with steroids within 1 week of study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Anticipated life expectancy of greater than 3 months
* Patients must have measurable disease either primary and/or metastatic masses reproducibly measurable in one or two diameters by Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 parameters by CT scan or MRI scan; positron emission tomography (PET) or octreotide scans are useful adjuncts but will not be used to measure response
* Granulocytes > 1,500/ml
* Platelets > 100,000/ml
* Hemoglobin >= 10 g/dl
* Creatinine < 1.5 x upper limit of normal (ULN) or creatinine clearance >= 50 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if liver metastases are present)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of veliparib, capecitabine and temozolomide administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be able to swallow pills

Exclusion Criteria:

* Prior chemotherapy with combination of capecitabine (or 5-flourouracil [5-FU]) "and" temozolomide (or dacarbazine [DTIC]) will be excluded; patients can have had prior therapies up to 3 prior chemotherapy regimens such as streptozocin, anthracyclines, irinotecan, etoposide, or a platinum agent including single agent capecitabine (or 5FU) or temozolomide (or DTIC).
* History of severe hypersensitivity reaction to capecitabine, 5-FU, temozolomide or DTIC will be excluded (i.e. anaphylaxis or anaphylactoid reactions)
* Patients who have active or uncontrolled infection or serious medical or psychiatric illness preventing informed consent or on intensive treatment
* Patients with brain metastases are excluded
* Patients with uncontrolled seizures or any neurological conditions resulting in increased risk for seizures are not eligible for study entry
* Patients with documented central nervous system (CNS) ischemia and/or infarction, whether symptomatic or discovered incidentally without clinical symptoms, will be excluded from study participation
* Patients with a history of the arterial or venous thromboembolism within =< 12 months of study entry are not eligible
* Human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy are excluded from the study
* Patients with another active malignancy within the past five years except for carcinoma in situ of cervix or in situ carcinoma of the bladder or non-melanomatous carcinoma of the skin
* Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities
* Patients who are receiving any other investigational agents
* Major surgical procedure within 4 weeks of treatment
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged QTc > 480 msec at baseline
  * Symptomatic congestive heart failure (CHF) of New York Heart Association (NYHA) functional class >= 3
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with capecitabine or temozolomide or veliparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose limiting toxicities defined as any toxicity in the first course evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 28 days

SECONDARY OUTCOMES:
Response rate measured as complete response, partial response or stable disease according to RECIST 1.1 criteria | 56 days (2 courses)
Response duration | Up to 4 weeks
Progression Free Survival | From start of treatment to time of progression or death, assessed up to 4 weeks
Overall Survival | Up to 4 weeks
Poly-adenosine diphosphate (ADP)-ribosylated (PAR) level | Baseline to day 15 of course 1

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided